CLINICAL TRIAL: NCT03143426
Title: Does 3D Visualisation Improve Performance of Laparoscopic Cholecystectomy by Junior Surgeons? A Randomised Controlled Trial
Brief Title: Does 3D Visualisation Improve Performance of Laparoscopic Cholecystectomy by Junior Surgeons?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Chea Chan Hooi, Doctor, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Complication Laparoscopic Cholecystectomy; Conversion Laparoscopic to Open Cholecystectomy
Keywords: 3D laparoscopic cholecystectomy; Junior surgeons; Complication; Conversion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D laparoscopic cholecystectomy (Experimental): Laparoscopic cholecystectomy will be performed under 3D visualisation.
  Interventions: Procedure: 3D laparoscopic cholecystectomy
- 2D laparoscopic cholecystectomy (No Intervention): Laparoscopic cholecystectomy will be performed under 2D visualisation, the standard viewing method used during all laparoscopic surgeries currently.

INTERVENTIONS:
Procedure: 3D laparoscopic cholecystectomy — Laparoscopic cholecystectomy will be performed under 3D visualization as opposed to 2D visualization (conventional method). 3D supposedly provide sharper view with better depth perception and therefore might lead to reduce complication rates.
  Arms: 3D laparoscopic cholecystectomy

SUMMARY:
Laparoscopic cholecystectomy (LC) is currently the most commonly performed major abdominal surgery in Western countries. Ever since the introduction of laparoscopic surgery in the late 1980s, cholecystectomies are now routinely performed laparoscopically; concomitantly the introduction and refinement of other laparoscopic abdominal surgeries have rapidly progressed due to the early experience and safety profile seen in LC.

The introduction of stereoscopes which allow for 3D visual feedback has been postulated to overcome setbacks encountered in conventional 2-dimensional (2D) laparoscopic surgery. Since its introduction in the mid-2000s, 3D visualisation has been proven to be advantageous over 2D visualisation, especially so within the context of training junior surgeons in controlled, experimental settings. The body of evidence on benefits of 3D visualisation within the clinical setting, i.e. when applied on live patients in operating theatres, remains small and weak. The previous publications however did not extrapolate any potential benefits on patients' well-being in correlation to their reported benefits and neither did they explore any potential benefits in reducing operative complications.

We decided to embark on a study to investigate any peri-operative advantage conferred on junior surgeons in performing LC using 3D visualisation as the majority of LCs in Sibu Hospital are carried out by junior surgeons.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is currently the most commonly performed major abdominal surgery in Western countries.1,2 Ever since the introduction of laparoscopic surgery in the late 1980s, cholecystectomies are now routinely performed laparoscopically; concomitantly the introduction and refinement of other laparoscopic abdominal surgeries have rapidly progressed due to the early experience and safety profile seen in LC.

Although the benefits of LC are well described (e.g. decreased post-operative pain, decreased need for post-operative analgesia, shortened hospital stay and earlier return to full activity),3,4 it is not completely risk-free. The surgeon's experience, or rather the lack of, has been previously identified as one of the significant correlations to inadvertent visceral injury.5 According to the European Association for Endoscopic Surgery, a minimum of 20 LCs are necessary before a surgeon is deemed able to perform it safely.6 This is consistent with the concept of the learning curve as analysed by Moore and Bennett; they noted that 90% of iatrogenic bile duct injuries occurred within the first 30 cases of the operating surgeon's experience.7 Publications on LC learning curve have identified the risk of an iatrogenic bile duct injury as 0.17% - 0.35% after a surgeon's 50th case as opposed to 1.3 - 1.7% when fewer than 50 cases.7,8 These higher risks of iatrogenic injuries have been attributed to the major setbacks encountered during conventional laparoscopic surgery, chiefly the lack of depth perception and tactile sensory feedback to the operating surgeon thus risking inadvertent injury to surrounding structures and imprecise dissection within the Calot's triangle. While the importance of senior supervision and guidance are indispensible, the technical short-comings of conventional laparoscopic surgery, i.e. the lack of depth perception, have led to the development of technology to allow for 3-dimensional (3D) visualisation.

The introduction of stereoscopes which allow for 3D visual feedback has been postulated to overcome these setbacks encountered in conventional 2-dimensional (2D) laparoscopic surgery. Since its introduction in the mid-2000s, 3D visualisation has been proven to be advantageous over 2D visualisation, especially so within the context of training junior surgeons in controlled, experimental settings.9,10 The body of evidence on benefits of 3D visualisation within the clinical setting, i.e. when applied on live patients in operating theatres, remains small and weak. These were mostly small, single-institution studies focused only on specific laparoscopic procedures such as hernia repair, distal gastrectomies,11 urologic12,13,14 and gynaecologic15,16 procedures.

Sakata and workers also believed that advantages conferred by 3D visualisation has been underreported and undermined by flawed study designs and utilised mostly earlier generation of 3D stereoscopes that has since been phased out, therefore undermining the clinical potential of 3D laparoscopy.17 Experience with utilisation of 3D visualisation in performing LC is still in its infancy and to the authors' knowledge, there have been no unfavourable results reported with the use of 3D visualisation for laparoscopic surgery. Data on direct comparison of 2D against 3D LC is still scarce; there are only three such studies and all demonstrated superiority of 3D over 2D visualisation in LC. These studies, though originating from tertiary institutions, are hampered by the limited numbers of patients operated using 3D visualisation (n = 8, 15 & 40 respectively).11,18,19 The third study,19 reported advantages of 3D visualisation conferred to junior surgeons in terms of reducing operative time, better depth perception and reduced subjective visual strain. The authors however did not extrapolate any potential benefits on patients' well-being in correlation to their reported benefits and neither did they explore any potential benefits in reducing operative complications.

Sibu Hospital is a 534-bedded tertiary and referral hospital for advanced specialised health care within the central region of Sarawak. Data from 2007 estimated that Sibu Hospital serves a population of at least 500 000 and this population is believed to have doubled to date.20 The department of general surgery is headed by a senior consultant surgeon (AD) and this department also serves as a training center for junior surgeons who have just completed their post-graduate qualifications. Under the tutelage of at least one senior consultant general surgeon, these junior surgeons are mentored through their early learning curves in performing major complicated surgeries, including LCs as it is the most common laparoscopic surgery being carried out in Sibu Hospital. Unpublished hospital data revealed that between 48 to 72 LCs are being performed annually since data collection began in 2010. Although major complications (e.g. adjacent organ injury) post-LC are rarely encountered in Sibu Hospital, relatively minor complications (e.g. excessive bleeding leading to prolonged theatre time) can still occur. In a bid to further reduce the complication rates of LC, we therefore decided to embark on a study to investigate any peri-operative advantage conferred on junior surgeons in performing LC using 3D visualisation as the majority of LCs in Sibu Hospital are carried out by junior surgeons.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled to undergo elective LC

Exclusion Criteria:

1. Patients below 18 years-old
2. Patients who declined to join the study
3. Patients with contraindications to undergo laparoscopic surgery (e.g. congestive cardiac failure, severe respiratory disease, uncorrected coagulopathy)
4. Patients with acute cholecystitis, gallbladder neck adherent to main biliary tree or dense omental adhesion to gallbladder
5. Patients with gallbladder tumour (suspected or confirmed)
6. Patients with variant biliary anatomy
7. Patients who had defaulted follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Complication rate | 6 months
  Intraoperative complications : Gallbladder perforation, adjacent organ injury, uncontrolled bleeding Post-operative : pain score, length of hospital stay, readmission, mortality

SECONDARY OUTCOMES:
Operative Time | 6 months
  Time taken between insertion of 4th port - cystic artery and cystic duct ligation - gallbladder full dissection.
Conversion to open cholecystectomy | 6 months
  To compare the rate of conversion between each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Hooi Chea, MS, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- Sibu Hospital, Sibu, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No